CLINICAL TRIAL: NCT05088343
Title: A Single-centre, Open, Single-dose, Self-control Study to Investigate the Effect of Hetrombopag on the Pharmacokinetics of Rosuvastatin in Healthy Chinese Adult Subjects.
Brief Title: Effect of Hetrombopag on the Pharmacokinetics of Rosuvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SHR8735-110
Record Dates: First submitted 2021-01-25; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Rosuvastatin Calcium; hetrombopag

STUDY DESIGN:
Intervention Model Description: rosuvastatin alone and then in combination with hetrombopag
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): rosuvastatin alone and then in combination with hetrombopag
  Interventions: Drug: Rosuvastatin; Drug: Hetrombopag

INTERVENTIONS:
Drug: Rosuvastatin — Single oral dose of rosuvastatin on Day 1 or co-administered with hetrombopag on Day 11.
Drug: Hetrombopag — 7.5 mg hetrombopag was administered on Day 6 to Day 11.

SUMMARY:
Effect of hetrombopag on the pharmacokinetics of rosuvastatin in healthy subjects.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effect of hetrombopag on pharmacokinetics of healthy Chinese adult subjects after oral administration of rosuvastatin calcium tablets. The secondary objective of the study is to evaluate the safety of rosuvastatin alone and when co-administered with hetrombopag.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
* Ability to complete the study as required by the protocol;
* Healthy male or female subjects aged 18 to 55 (including 18 and 55) at the date of signing the informed consent;
* Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26).

Exclusion Criteria:

* Allergic constitution;
* History of drug use, or drug abuse screening positive;
* Alcoholic or often drinkers;
* History of deep vein thrombosis, or any other thromboembolic event;
* A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
* Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 0-72 hours post dose
Area Under the plasma concentration vs time curve (AUC0-72) | 0-72 hours post dose
Area under the blood concentration vs time curve (AUC0-inf) | 0-infinity

SECONDARY OUTCOMES:
Other pharmacokinetics parameters of rosuvastatin | 0-72 hours post dose
  Tmax
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Ding, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xueying General Ding, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided